CLINICAL TRIAL: NCT04475692
Title: A Multicentre Pilot Randomised Control Trial of an Adapted Mobile Rehabilitation System for Self-directed Rehabilitation and Improved Upper Limb Outcomes in Stroke Survivors With Upper Limb Weakness
Brief Title: Self-directed Adapted Gaming Exercises for Stroke Survivors
Acronym: SAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20CX5959
Record Dates: First submitted 2020-07-09; First posted 2020-07-17 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Cerebrovascular Accident
Keywords: Rehabilitation; Upper limb; Technology; Self-administered; Self-directed
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: A multicentre pilot RCT, parallel design, comparing intervention group (self-selected dose of self-directed technology-based UL exercise as an adjunct to conventional care) with a control group receiving conventional care only.
Who Masked: Outcomes Assessor
Masking Description: This will be an assessor-blinded protocol, due to the nature of the intervention, participants cannot be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Conventional care will continue.
  Participants (and proxy, where relevant) will be trained to use the intervention platform (GripAble). Participants will be loaned a GripAble device and advised to continue a self-selected training dose throughout the intervention period.
  Weekly follow-up phone calls will be conducted, remote tech support will be available. Adherence with the intervention will be remotely monitored via an inbuilt data capture system.
  At 3months post stroke, the intervention period will conclude, outcome measures will be implemented. Participants will be invited to complete a post intervention survey and interview. A purposive sample of participants will be invited to participate in an UL activity monitoring sub-study.
  At 6months post stroke, follow-up outcome measures will be implemented. Participants will be invited to take part in a research implementation feedback survey.
  Interventions: Behavioral: Repetitive, task-specific upper limb practice; Other: Conventional care
- Control (Active Comparator): Baseline data collection and outcome measures will be completed.
  Conventional care will continue, no restrictions/specifications will be placed on this.
  At 3months post stroke, UL outcome measures will be implemented. A purposive sample of participants will be invited to participate in an UL activity monitoring sub-study.
  At 6months post stroke, follow-up UL outcome measures will be implemented. Participants will be invited to take part in a research implementation feedback survey.
  Interventions: Other: Conventional care

INTERVENTIONS:
Behavioral: Repetitive, task-specific upper limb practice — A self-directed upper limb intervention (implementing a self-selected dose). This intervention uses an adapted upper limb rehabilitation system to support repetitive upper limb training for stroke survivors.
  Other Names: Gamified exercise; Interactive gaming; Virtual reality; Self-directed upper limb rehabilitation
  Arms: Intervention
Other: Conventional care — Conventional care is the standard care offered to stroke patients in their respective settings. In this context it is guided by Royal College of Physicians (2016). For the purposes of this work, conventional care encompasses any rehabilitation or support services accessed by participants within the primary or secondary care setting, including private therapy services, charity-led exercise groups etc. Conventional care will not be specified in the context of this work, as it is complex in nature and varies between settings.

SUMMARY:
A pilot multicentre randomised control trial (RCT), examining upper limb (UL) outcomes amongst stroke survivors implementing a technology-based, self-directed UL intervention as an adjunct to conventional care.

DETAILED DESCRIPTION:
Title: A multicentre pilot randomised control trial (RCT) of an adapted mobile rehabilitation system (GripAble) for self-directed upper limb (UL) rehabilitation and improved UL outcomes in stroke survivors with UL weakness.

Design: Interventional (clinical trial). A multicentre pilot RCT, parallel design, comparing intervention group (self-selected dose of self-directed technology-based UL exercise as an adjunct to conventional care) with a control group receiving conventional care only. A mixed methods research design will be implemented. This will be an assessor-blinded protocol, due to the nature of the intervention, participants cannot be blinded. This will be an internal pilot, if no changes are made to the protocol and additional funding is secured, the data from this pilot work will be used be used as part of an adequately powered RCT.

Aims: To test research design considerations in preparation for a definitive multicentre RCT. To explore the hypothesis that stroke survivors with UL weakness will engage in self-directed exercise (without direct professional supervision) as an adjunct to conventional care and demonstrate significant improvement in UL outcomes when provided with an adapted mobile rehabilitation system, compared with a control group participating in conventional care only.

Outcome Measures: The primary end point outcome will be based on intention to treat analysis on the Fugl Meyer Upper Extremity Assessment (FM-UE) at 6months post randomisation, controlled for baseline.

Additional/ secondary outcome measures will include: The Action Arm Research Test (ARAT), Apple watch activity monitors (implementing tailor-made machine learning methods to interpret UL movement data), Barthel Index (BI), Modified Rankin Scale (mRS), Hospital Anxiety and Depression Scale (HADS), Faces Pain Rating Scale (FPRS), Stanford Fatigue Visual Numeric Scale (SFVNS).

Assessments administered for the purpose of sample description (sub group analysis) and stratification will include: National Institutes of Health Stroke Scale (NIHSS), Edinburgh Handedness Scale (EHS), Montreal Cognitive Assessment (MOCA), Likert scale participant feedback forms (devised for the purposes of the current study). For purposively sampled sub-groups of participants, sub studies will explore bilateral naturalistic UL activity patterns in free living (intervention and control groups) and qualitative interviews will examine the mechanisms of behavioral change as relevant to the intervention (intervention group only).

Population: A convenience sample of 72 stroke survivors will be screened and consented by delegated health care practitioners (HCPs) or researchers at participating sites (i.e Co-Investigators (Co-Is)). Co-Is will also be invited to complete end-point feedback forms.

Eligibility: Participants will be 18yrs or over, acute/sub-acute stroke survivors with new UL impairment, fitting inclusion criteria specified herewith.

Duration: Participants' enrolment in the study will last up to 6months. The study recruitment phase will open for a total of 12months. The overall research period, including analysis and write up is anticipated to last 21months.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive status that would permit for use /supported use of intervention device and engagement in protocol related trainings/assessment. To be indicated by treating clinician at point of screening, formal capacity assessment to be conducted as/if appropriate. Easy read patient information sheet (PIS) and training materials will be implemented to support patients presenting with specific cognitive and/or communication needs.
* Stroke diagnosis (can be first or subsequent stroke, unilateral haemorrhagic or ischemic) 4 weeks max post stroke at time of recruitment.
* Can communicate in English, that is, sufficient for completion of intervention and outcome measures. It is advisable that a decision to include or exclude those with significant expressive or receptive communication impairment should be made following consultation with the treating speech and language therapist (SLT) to ensure all reasonable accommodations are made to support participation.
* UL motor deficit post stroke (bilateral/unilateral) (according to National Institutes of Health Stroke Score (NIHSS) item 5), distal UL power >1 /5 on the Oxford Rating Scale (Medical Research Council Manual Muscle Testing scale) or voluntary finger extension of the thumb and/or two or more fingers of the affected hand (to 10° or more). The presence of sensory impairment (including neglect syndrome) or movement disorder (apraxia) is not a contraindication to enrolment as long as there is a concurrent motor deficit (as described above).

Exclusion Criteria:

* Patients already enrolled an interventional neuro rehabilitation trial.
* Patients enrolled in clinical trials that contraindicate co-enrolment.
* Patients presenting with unstable medical conditions/medical contraindications as determined by treating medical consultant (these patients may be approached at a later date should their condition improve).
* Patients with uncontrolled photosensitive epilepsy/Other neurological symptoms that may be exacerbated by required focus on light emitting diode (LED) screen/moving object on screen).
* Those registered blind/with uncompensated/uncorrected visual deficits.
* Behavioural/affective dysfunction which could influence the ability of the person to engage with the research protocol and/or pose risk to the participating researchers (in circumstances such as follow-up community visits).
* Other concomitant neurological disorders affecting upper extremity motor function (Multiple Sclerosis, Spinal Cord Injury, Brachial Plexus or Radial Nerve Injury).
* Unremitting arm pain at rest.
* Pre-existing UL impairment with known and significant disruption to range of motion, motor or functional performance (fracture, arthritic changes, other known musculoskeletal problems).
* Skin condition apparent on the ventral UE such that might place participant at risk of irritation in the context of repeated physical contact (such as that associated with the intervention).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment- Upper Extremity (FM-UE) | Change between scores from baseline (0-1month post stroke) to 3months post stroke and 6months post stroke
  Upper limb (UL) impairment-based measure: The FM-UE assesses UL impairment in terms of synergistic motor control. It has 3 categories, comprised of 22 sub questions scored on a 3-point ordinal scale (0=unable, 1=partial, 2=near normal). The sum of the categories ranges between 0 and 66 points (66 = normal function). The FM-UE has shown excellent inter-rater reliability (Sullivan et al., 2011)(Duncan, Goldstein, Matchar, Divine, & Feussner, 1992) moderate to good responsiveness (Lundquist & Maribo, 2017) and good concurrent validity when compared with similar tests of arm motor functioning.

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) | Change between scores from baseline (0-1month post stroke) to 3months post stroke and 6months post stroke
  The ARAT is an UL capacity test which assesses the ability to grasp, move and release objects of various sizes, weights and shapes. It has 19 sub questions scored on a 4-point ordinal scale, adding up to a total score between 0 and 57 points (57 = normal capacity).

CONTACTS AND LOCATIONS:
Overall Officials: Jane Burridge, Study Chair — University of Southampton
Locations (1):
- Paul Bentley, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be used for the specified purposes only. Data will not be shared outside of the primary research team.

REFERENCES:
- [Derived] Broderick M, Burridge J, Demain S, Johnson L, Brereton J, O'Shea R, Bentley P. Multicentre pilot randomised control trial of a self-directed exergaming intervention for poststroke upper limb rehabilitation: research protocol. BMJ Open. 2024 Jan 19;14(1):e077121. doi: 10.1136/bmjopen-2023-077121. PMID 38245014